CLINICAL TRIAL: NCT05855733
Title: Radiofrequency Treatment for Pilonidal Disease : Clinical Investigation on Safety of Use, Efficacy and Patient Satisfaction at 6 Months
Brief Title: Radiofrequency Treatment for Pilonidal Disease : Safety of Use, Efficacy and Patient Satisfaction at 6 Months
Acronym: RaTPiD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RaTPiD
Record Dates: First submitted 2023-04-17; First posted 2023-05-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Infected Pilonidal Sinus
Keywords: Radiofrequency
MeSH Terms: interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency (Experimental): treatment of pilonidal disease according to the Fistura procedure
  Interventions: Device: radiofrequency treatment

INTERVENTIONS:
Device: radiofrequency treatment — patient undergoing radiofrequency using the Fistura procedure for treatment of a infected pilonidal sinus

SUMMARY:
Infected pilonidal sinus is a common suppuration that occurs twice as often in men as in women, usually between the ages of 15 and 30. Clinical diagnosis is easy, whether the presentation is acute or chronic. Exeresis with a wound left open requiring secondary postoperative healing is the most widely practiced technique in France because its recurrence rate is the lowest, but it has the disadvantage of requiring daily or even twice-daily local nursing care, long healing, and a break in activity.

In order to limit the disadvantages of the open technique, "conservative" minimally invasive techniques have also recently been developed in response to strong patient demand: such as endoscopic treatment (EPSIT = Endoscopic Pilonidal Sinus Treatment, or VAAPS = Video-Assisted Ablation of Pilonidal Sinus), or the SiLaT (Sinus Laser Therapy) laser.

More recently, radiofrequency has emerged as a new technique in the treatment of hemorrhoidal pathology according to the Rafaelo procedure as well as the Fistura procedure for anal fistulas. The principle of the treatment is similar to that of the laser, based on radio frequency thermocoagulation using very high frequency electromagnetic waves (4MHz), similar to the principle of microwaves. However, its use in the infected pilonidal sinus has not yet been described. The fibers used in anal fistulas are perfectly adapted to the treatment of the pilonidal sinus. In addition, and in contrast to the laser, several fiber diameters are available depending on the size of the fistula path(s). For example, the large diameters of 9 Fr seem to be more adapted to the deep and wide cavities of the pilonidal sinuses than those of the SiLaT, which has a single fiber diameter. The investigators can therefore think that this type of fibers could allow a more efficient destruction of the granulation tissues and a better docking of the cavity walls.

According to published studies in the treatment of anal fistulas, the safety profile of this treatment is perfectly reassuring since the penetrance of the energy released does not exceed 3 mm in depth.

The aim of this study is to propose a competing alternative to the SiLaT laser, which is radiofrequency according to the Fistura® procedure, by evaluating its safety, efficacy and patient satisfaction on a series of consecutive patients treated

ELIGIBILITY:
Inclusion Criteria:

* patient presenting an infected pilonidal sinus requiring an surgical procedure, at the exception of acute abscess stage
* Patient aged 18 or above
* For Women Of Child Bearing Age, use of efficient contraceptive (less than 1% failure)
* Patient with health insurance coverage
* French-speaking patient
* Signed written informed consent

Exclusion Criteria:

* Patient already included in a type 1 interventional research protocol (RIPH1)
* Patient with cardiac disease (including pacemaker)
* Patient with skin infection
* Patient for whom local or general anesthesia is contraindicated
* patient presenting an anal infectious disease, or an anal fissure or who have previously had a stapled hemorrhoidopexy (Longo procedure) with metallic staples.
* Patient using anticoagulant or anti-platelet agent (at the exception of aspirin)
* Patient suffering from innate hemostasis and/or coagulation disorder
* Patient for whom MRI is contraindicated
* Pregnant or Breastfeeding women
* Patient under guardianship or curatorship
* Patient incarcerated
* Patient under legal protection
* Patient refusing follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of at least one complication of the surgery | Within 15days after surgery
  incidence rate of haemorrhagic complication or acute urinary retention or other complication (such as post surgery abcess, localized infection, haematoma)

SECONDARY OUTCOMES:
Incidence rate of of haemorrhagic complication after surgery | Within 15days after surgery
Incidence rate of acute urinary retention after surgery | Within 15days after surgery
Incidence rate of other complication of surgery | Within 15days after surgery
  incidence rate of other complication such as post surgery abcess, localized infection, haematoma
Evaluation of post-surgery pain | within 15 days post surgery
  Patient will be asked daily to evaluate post surgery pain using a Numerical Rating Scale (NRS). Patients will be asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero represents 'no pain at all' whereas10 represents 'the worst pain ever possible'.
Evaluation of radiofrequency treatment efficiency | 6 months after surgery
  During the last patient visit, a clinical evaluation will be performed during which closure of all existing fistula external opening will be assessed (Yes or No), as well as the absence or presence of abcess and new external opening (Yes or no) . The patient will be asked to evaluate the presence or absence of pain (yes or no)
  The Treatment will be evaluated as efficient if there is closure of all fistula external opening AND absence of pain AND absence of abscess or new external opening
Length of the medical leave after surgery | within 6 months post surgery
  Record of number of medical leave days prescribed after surgery Record of number of day after surgery necessary before returning to normal activity.
Measurement of patient satisfaction after surgery | 1 month and 6 months post surgery
  patient will evaluate their satisfaction regarding their surgery using a visual 5 point scale ranking from "very unsatified" to "very satisfied"

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Velotti N, Manigrasso M, Di Lauro K, Araimo E, Calculli F, Vertaldi S, Anoldo P, Aprea G, Simone G, Vitiello A, Musella M, Milone M, De Palma GD, Milone F, Sosa Fernandez LM. Minimally Invasive Pilonidal Sinus Treatment: A Narrative Review. Open Med (Wars). 2019 Aug 7;14:532-536. doi: 10.1515/med-2019-0059. eCollection 2019. PMID 31428682
- [Background] Romic I, Augustin G, Bogdanic B, Bruketa T, Moric T. Laser treatment of pilonidal disease: a systematic review. Lasers Med Sci. 2022 Mar;37(2):723-732. doi: 10.1007/s10103-021-03379-x. Epub 2021 Jul 22. PMID 34291332
- [Background] Meinero P, Mori L, Gasloli G. Endoscopic pilonidal sinus treatment (E.P.Si.T.). Tech Coloproctol. 2014 Apr;18(4):389-92. doi: 10.1007/s10151-013-1016-9. Epub 2013 May 17. PMID 23681300
- [Background] Keogh KM, Smart NJ. The proposed use of radiofrequency ablation for the treatment of fistula-in-ano. Med Hypotheses. 2016 Jan;86:39-42. doi: 10.1016/j.mehy.2015.11.019. Epub 2015 Nov 26. PMID 26804594
- [Background] Eddama MMR, Everson M, Renshaw S, Taj T, Boulton R, Crosbie J, Cohen CR. Radiofrequency ablation for the treatment of haemorrhoidal disease: a minimally invasive and effective treatment modality. Tech Coloproctol. 2019 Aug;23(8):769-774. doi: 10.1007/s10151-019-02054-2. Epub 2019 Aug 9. PMID 31399891